CLINICAL TRIAL: NCT04868890
Title: A Randomized, Double-Blinded, Placebo-Controlled Phase II Study to Evaluate the Safety and Efficacy of Inhaled Ampion in Adults With Respiratory Distress Due to COVID-19
Brief Title: A Study of Inhaled Ampion in Adults With Respiratory Distress Due to COVID-19
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The AP-019 study was prematurely terminated by the sponsor after determining that insufficient events were occurring to analyze the primary endpoint.
Sponsor: Ampio Pharmaceuticals. Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AP-019
Record Dates: First submitted 2021-04-22; First posted 2021-05-03 (Actual); Results first posted 2022-12-07 (Actual); Last update posted 2022-12-07 (Actual); Status verified 2022-05

CONDITIONS: Covid19
MeSH Terms: conditions — COVID-19 | interventions — aspartyl-alanyl-diketopiperazine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Active (Experimental): Ampion
  Interventions: Biological: Ampion
- Control (Placebo Comparator): Placebo
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: Ampion — Inhaled Ampion
  Arms: Active
Other: Placebo — Inhaled Placebo
  Arms: Control

SUMMARY:
This is phase II study to evaluate the safety and efficacy of inhaled Ampion in adults with respiratory distress due to COVID-19

DETAILED DESCRIPTION:
The severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) has resulted in the pandemic spread of coronavirus disease 2019 (COVID-19), which has a high rate of infection, has a high rate of hospitalization, has overwhelmed healthcare systems, and can be fatal.

Ampion is the low molecular weight filtrate of human serum albumin with the in vitro ability to modulate inflammatory cytokine levels. Ampion has the potential to improve clinical outcomes for COVID-19 patients by reducing inflammatory cytokines correlated with the disease and respiratory complications, such as Acute Lung Injury (ALI) and Acute Respiratory Distress Syndrome (ARDS).

This study aims to evaluate the effects of Ampion on mortality and clinical outcomes in patients with respiratory distress due to COVID-19.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, ≥ 18 years old
2. Diagnosed with COVID-19, as evaluated by laboratory diagnostic test or diagnosis based on radiological clinical findings.
3. Baseline severity categorization of severe or critical COVID-19 infection per FDA Guidance for developing drugs and biological products for COVID-19 (February 2021):

   1. Severe COVID-19:

      * Symptoms suggestive of severe systemic illness with COVID-19, which could include shortness of breath or respiratory distress
      * Clinical signs indicative of severe systemic illness with COVID-19, such as respiratory rate ≥ 30 per minute, heart rate ≥ 125 per minute, SpO2 ≤ 93% on room air at or PaO2/FiO2 < 300
   2. Critical COVID-19:

      * Oxygen delivered by high-flow nasal cannula (heated, humidified, oxygen delivered via reinforced cannula at flow rates > 20 L/min with fraction of oxygen ≥ 0.5) or
      * Non-invasive mechanical or endotracheal mechanical ventilation
4. Informed consent obtained from the patient or the patient's legal representative.

Exclusion Criteria:

1. As a result of the medical review and screening investigation, the Principal Investigator considers the patient unfit for the study and/or progression to death is imminent and inevitable irrespective of the provision of treatments.
2. Clinical diagnosis of respiratory failure requiring ECMO and/or therapy is not available due to limitation.
3. Shock defined by systolic blood pressure <90 mm Hg, or diastolic blood pressure <60 mm Hg or requiring vasopressors.
4. Multi-organ dysfunction/failure.
5. Patient has severe chronic obstructive or restrictive pulmonary disease (COPD) (as defined by prior pulmonary function tests), chronic renal failure, or significant liver abnormality (e.g., cirrhosis, transplant, etc.).
6. Patient has chronic conditions requiring chemotherapy or immunosuppressive medication.
7. A history of allergic reactions to human albumin (reaction to non-human albumin such as egg albumin is not an exclusion criterion) or ingredients in 5% human albumin (N- acetyltryptophan, sodium caprylate).
8. Prolonged QT interval.
9. Patient has known pregnancy or is currently breastfeeding.
10. Patient planning to become pregnant, or father a child, during the treatment and follow-up period and/or is not willing to remain abstinent or use contraception.
11. Participation in another clinical trial (not including treatments for COVID-19 as approved by the FDA through expanded access, emergency, or compassionate use), or participation in a trial such that enrollment in this study would fall within the time frame of the half-life of the other investigational product(s).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2021-06-22 (Actual); Primary Completion 2022-02-16 (Actual); Study Completion 2022-04-13 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Ampio Pharmaceuticals, Englewood, Colorado, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Active: Ampion
  Ampion: Inhaled Ampion (8mL) administered four times daily for 5 days
- Control: Placebo
  Placebo: Inhaled Placebo (8mL) administered four times daily for 5 days
Period: Overall Study
Arm/Group | Active | Control
Started | 64 | 65
Completed | 61 | 59
Not Completed | 3 | 6
Not completed — Death | 2 | 1
Not completed — Withdrawal by Subject | 1 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Active | Control | Total
Number analyzed (Participants) | 64 | 65 | 129
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.9 (15.2) | 56.9 (16.6) | 54.9 (16.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21 | 26 | 47
  Male | 43 | 39 | 82
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 24 | 26 | 50
  Not Hispanic or Latino | 40 | 39 | 79
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 36 | 33 | 69
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 3 | 5
  White | 26 | 29 | 55
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 28 | 32 | 60
  India | 36 | 33 | 69
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 29.4 (7.1) | 28.5 (5.4) | 28.9 (6.3)

OUTCOME MEASURES:

1. Primary Outcome: Clinical Improvement of Participants of Ampion Compared to Placebo
Description: Change in ordinal scale from baseline through Day 5 and through Day 28. The WHO's 8 point ordinal scale reflects the highest level of support the subject required on the day being recorded. 0 = No clinical or virological evidence of infection; 1 = no limitation of activities; 2 = limitation of activities; 3 = Hospitalized, no oxygen; 4 = Hospitalized, oxygen by mask or nasal prongs; 5 = Hospitalized, non-invasive ventilation or high-flow oxygen, 6 = Hospitalized, mechanical ventilation; 7 = Hospitalized, ventilation + additional organ support - pressors, RRT, ECMO; 8 = Death. A negative difference in mean score constitutes a reduction in the severity of clinical intervention.
Time Frame: Day 28
Population: Intent to Treat (ITT)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Active | Control
Number analyzed (Participants) | 64 | 65
score on a scale
  Day 5 | -0.5 (0.95) | -0.4 (0.73)
  Day 28 | -4.1 (0.63) | -4.0 (0.49)

2. Secondary Outcome: The Number of Participants With Treatment Emergent Adverse Events of Ampion Compared to Placebo
Description: Number of subjects with treatment emergent adverse events (TEAEs) and serious adverse events (SAEs) of treatment of inhalation Ampion compared to Placebo. AEs were assessed based on symptoms as a severity rating of mild, moderate, or severe. The relationship between AE and study drug was determined as either unrelated, possibly related, or related. SAEs are defined as resulting death, life threatening, requires prolonged hospitalization, results in persistent or significant disability/incapacity, or results in congenital anomaly/birth defect.
Time Frame: Day 60
Population: Safety
Measure: Count of Participants; unit: Participants
Arm/Group | Active | Control
Number analyzed (Participants) | 64 | 65
Participants
  Treatment Emergent Adverse Events (TEAE's) | 21 | 18
  Study Drug Related TEAE's | 0 | 1
  Moderate or Severe TEAE's | 10 | 11
  Serious Adverse Events (SAE's) | 2 | 4

ADVERSE EVENTS:
Time Frame: Day 60
Description: Patients were followed for the occurrence of Adverse Events for 60 days following the first dose of study medication.
Arm/Group | Active | Control
All-Cause Mortality (participants affected / at risk) | 2/64 | 1/65
Serious Adverse Events (participants affected / at risk) | 2/64 | 4/65
Other Adverse Events (participants affected / at risk) | 21/64 | 18/65
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Active (N=64) | Control (N=65)
Chest Pain (General disorders) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 0 (0) | 1 (1)
Acute Respiratory Distress Syndrome (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Active (N=64) | Control (N=65)
Abdominal Discomfort (Gastrointestinal disorders) | 2 (2) | 0 (0)
Constipation (Gastrointestinal disorders) | 2 (2) | 1 (1)
Asthenia (General disorders) | 2 (2) | 2 (2)
Fatigue (General disorders) | 4 (4) | 1 (1)
Pain (General disorders) | 2 (2) | 2 (2)
Pyrexia (General disorders) | 3 (3) | 1 (1)
Alanine Aminotransferase Increased (Investigations) | 1 (1) | 2 (2)
Blood Lactate Dehydrogenase Increased (Investigations) | 2 (2) | 0 (0)
Blood Urea Abnormal (Investigations) | 3 (3) | 3 (3)
C-Reactive Protein Increased (Investigations) | 2 (2) | 0 (0)
Platelet Count Abnormal (Investigations) | 2 (2) | 0 (0)
Serum Ferritin Increased (Investigations) | 2 (2) | 0 (0)
Headache (Nervous system disorders) | 3 (3) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Aspartate Aminotransferase Increased (Investigations) | 1 (1) | 0 (0)
Blood Bicarbonate Abnormal (Investigations) | 0 (0) | 1 (1)
Blood Creatine Abnormal (Investigations) | 1 (1) | 0 (0)
Blood Creatine Increased (Investigations) | 1 (1) | 0 (0)
Blood Potassium Abnormal (Investigations) | 1 (1) | 1 (1)
Blood Sodium Abnormal (Investigations) | 0 (0) | 1 (1)
Electrocardiogram QT Prolonged (Investigations) | 0 (0) | 1 (1)
Lymphocyte Count Decreased (Investigations) | 1 (1) | 0 (0)
Neutrophil Count Increased (Investigations) | 1 (1) | 0 (0)
White Blood Cell Count Abnormal (Investigations) | 0 (0) | 1 (1)
White Blood Cell Count Increased (Investigations) | 1 (1) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Type 2 Diabetes Mellitus (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Musculoskeletal Chest Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Memory Impairment (Nervous system disorders) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 1 (1)
Haematuria (Renal and urinary disorders) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Nasal Discomfort (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Orthopnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
The AP-019 study was prematurely terminated by the sponsor after determining that insufficient events were occurring to analyze the primary endpoint.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2022-03-18): https://cdn.clinicaltrials.gov/large-docs/90/NCT04868890/Prot_000.pdf
  • Statistical Analysis Plan (2022-08-11): https://cdn.clinicaltrials.gov/large-docs/90/NCT04868890/SAP_001.pdf